CLINICAL TRIAL: NCT01831050
Title: A Phase 4, Randomized Study to Evaluate the Safety and the Humoral and Intestinal Immunogenicity of One or Two Additional Doses of Licensed Inactivated Polio Vaccines (IPVs) in Latin American Infants Previously Vaccinated With Bivalent Oral Polio Vaccines (bOPVs)
Brief Title: Safety and Immunogenicity of 1 or 2 Doses of IPV in Latin American Infants Primed With Bivalent OPV Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fidec Corporation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 12-1460
Record Dates: First submitted 2013-04-10; First posted 2013-04-15 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Poliomyelitis
Keywords: Poliovirus; Inactivated poliovirus vaccine; Trivalent oral polio vaccine; Bivalent oral polio vaccine; Stool shedding index; Polio eradication
MeSH Terms: conditions — Poliomyelitis | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- G1: Sanofi bOPV Control (Experimental): 210 infants receiving Bivalent Oral Polio Vaccine (bOPV) at 6, 10 and 14 weeks with Monovalent Oral Polio Vaccine Type 2 (mOPV2) challenge at 18 weeks
  Interventions: Biological: Bivalent Oral Polio Vaccine (bOPV); Biological: Monovalent Oral Polio Vaccine Type 2 (mOPV2)
- G2: Sanofi bOPV Control (Experimental): 210 infants receiving Bivalent Oral Polio Vaccine (bOPV) at 6, 10 and 14 weeks with Monovalent Oral Polio Vaccine Type 2 (mOPV2) challenge at 40 weeks
  Interventions: Biological: Bivalent Oral Polio Vaccine (bOPV); Biological: Monovalent Oral Polio Vaccine Type 2 (mOPV2)
- G3: Trivalent OPV Control (Experimental): 100 infants receiving Trivalent Oral Polio Vaccine (tOPV)' at 6, 10 and 14 weeks with Monovalent Oral Polio Vaccine Type 2 (mOPV2) challenge at 18 weeks
  Interventions: Biological: Trivalent Oral Polio Vaccine (tOPV); Biological: Monovalent Oral Polio Vaccine Type 2 (mOPV2)
- G4: Sanofi bOPV, Sanofi IPV (Experimental): 210 infants receiving Bivalent Oral Polio Vaccine (bOPV) at 6, 10 and 14 weeks and 1 dose of Sanofi-Pasteur IPV (Sanofi IPV) at 14 weeks with Monovalent Oral Polio Vaccine Type 2 (mOPV2) challenge at 18 weeks
  Interventions: Biological: Bivalent Oral Polio Vaccine (bOPV); Biological: Monovalent Oral Polio Vaccine Type 2 (mOPV2); Biological: Sanofi-Pasteur IPV (Sanofi IPV)
- G5: Sanofi bOPV, Sanofi 2 IPV (Experimental): 210 infants receiving Bivalent Oral Polio Vaccine (bOPV) at 6, 10 and 14 weeks and 2 dose of Sanofi-Pasteur IPV (Sanofi IPV) at 14 and 36 weeks with Monovalent Oral Polio Vaccine Type 2 (mOPV2) challenge at 40 weeks
  Interventions: Biological: Bivalent Oral Polio Vaccine (bOPV); Biological: Monovalent Oral Polio Vaccine Type 2 (mOPV2); Biological: Sanofi-Pasteur IPV (Sanofi IPV)
- G6: Sanofi bOPV, GSK IPV (Experimental): 50 infants receiving Bivalent Oral Polio Vaccine (bOPV) at 6, 10 and 14 weeks and 1 dose of Glaxo SmithKline IPV (GSK IPV) at 14 weeks with Monovalent Oral Polio Vaccine Type 2 (mOPV2) challenge at 18 weeks
  Interventions: Biological: Bivalent Oral Polio Vaccine (bOPV); Biological: Monovalent Oral Polio Vaccine Type 2 (mOPV2); Biological: Glaxo SmithKline IPV (GSK IPV)
- G7: Sanofi bOPV, GSK 2 IPV (Experimental): 190 infants receiving Bivalent Oral Polio Vaccine (bOPV) at 6, 10 and 14 weeks and 2 doses of Glaxo SmithKline IPV (GSK IPV) at 14 and 36 weeks with Monovalent Oral Polio Vaccine Type 2 (mOPV2) challenge at 40 weeks
  Interventions: Biological: Bivalent Oral Polio Vaccine (bOPV); Biological: Monovalent Oral Polio Vaccine Type 2 (mOPV2); Biological: Glaxo SmithKline IPV (GSK IPV)
- G8: Sanofi bOPV, SII IPV (Experimental): 50 infants receiving Bivalent Oral Polio Vaccine (bOPV) at 6, 10 and 14 weeks and 1 dose of Serum Institute of India IPV (SII IPV) at 14 weeks with Monovalent Oral Polio Vaccine Type 2 (mOPV2) challenge at 18 weeks
  Interventions: Biological: Bivalent Oral Polio Vaccine (bOPV); Biological: Monovalent Oral Polio Vaccine Type 2 (mOPV2); Biological: Serum Institute of India IPV (SII IPV)
- G9: Sanofi bOPV, SII 2 IPV (Experimental): 190 infants receiving Bivalent Oral Polio Vaccine (bOPV) at 6, 10 and 14 weeks and 2 doses of Serum Institute of India IPV (SII IPV) at 14 and 36 weeks with Monovalent Oral Polio Vaccine Type 2 (mOPV2) challenge at 40 weeks
  Interventions: Biological: Bivalent Oral Polio Vaccine (bOPV); Biological: Monovalent Oral Polio Vaccine Type 2 (mOPV2); Biological: Serum Institute of India IPV (SII IPV)

INTERVENTIONS:
Biological: Bivalent Oral Polio Vaccine (bOPV) — Produced by Sanofi Pasteur, Lyon, France, bivalent OPV vaccine contains types 1 and 3 polioviruses and it is indicated for supplementary immunization activities in children from 0 to 5 years of age to prevent or contain outbreaks caused by these 2 serotypes.
  Other Names: Bivalent Oral Polio Vaccine; bOPV
  Arms: G1: Sanofi bOPV Control; G2: Sanofi bOPV Control; G4: Sanofi bOPV, Sanofi IPV; G5: Sanofi bOPV, Sanofi 2 IPV; G6: Sanofi bOPV, GSK IPV; G7: Sanofi bOPV, GSK 2 IPV; G8: Sanofi bOPV, SII IPV; G9: Sanofi bOPV, SII 2 IPV
Biological: Trivalent Oral Polio Vaccine (tOPV) — Produced by Sanofi Pasteur, Lyon, France, trivalent OPV vaccine contains types 1, 2, and 3 polioviruses and it is indicated for routine and supplementary prevention of poliomyelitis in children from 0 to 5 years of age.
  Other Names: "OPVERO"; Trivalent Oral Polio Vaccine; tOPV
  Arms: G3: Trivalent OPV Control
Biological: Monovalent Oral Polio Vaccine Type 2 (mOPV2) — Licensed monovalent OPV type 2 vaccine (mOPV2) by Glaxo SmithKline, Rixensart, Belgium. Polio Sabin Mono Two (oral) is a monovalent, live attenuated poliomyelitis virus vaccine of the Sabin strain Type 2 (P 712, Ch, 2ab), propagated in MRC5 human diploid cells.
  Other Names: Polio Sabin Mono Two; Monovalent Oral Polio Vaccine Type 2; mOPV2
Biological: Sanofi-Pasteur IPV (Sanofi IPV) — Inactivated poliovirus vaccine is produced by Sanofi-Pasteur as a sterile suspension of 3 types of poliovirus. Each dose of vaccine (0.5 mL) contains 40 D antigen units of Mahoney strain (Type 1); 8 D antigen units of MEF-1 strain (Type 2); and 32 D antigen units of Saukett strain (Type 3).
  Other Names: Sanofi-Pasteur IPV; IPOL; IMOVAX; Sanofi IPV
  Arms: G4: Sanofi bOPV, Sanofi IPV; G5: Sanofi bOPV, Sanofi 2 IPV
Biological: Glaxo SmithKline IPV (GSK IPV) — Inactivated poliovirus vaccine is produced by Glaxo SmithKline, Rixensart, Belgium, as a sterile suspension of 3 types of poliovirus. Each dose of vaccine (0.5 mL) contains 40 D antigen units of Mahoney strain (Type 1); 8 D antigen units of MEF-1 strain (Type 2); and 32 D antigen units of Saukett strain (Type 3).
  Other Names: Glaxo SmithKline IPV; POLIORIX; (GSK IPV)
  Arms: G6: Sanofi bOPV, GSK IPV; G7: Sanofi bOPV, GSK 2 IPV
Biological: Serum Institute of India IPV (SII IPV) — Inactivated poliovirus vaccine produced by Nederland's Vaccin Instituut in Bilthoven, The Netherlands (acquired recently by Serum Institute of India [SII]) is licensed in the producing country and prequalified by the WHO. It consists of a sterile suspension of 3 types of poliovirus. Each dose of vaccine (0.5 mL) contains 40 D antigen units of Mahoney strain (Type 1); 8 D antigen units of MEF-1 strain (Type 2); and 32 D antigen units of Saukett strain (Type 3).
  Other Names: Serum Institute of India IPV; SII IPV
  Arms: G8: Sanofi bOPV, SII IPV; G9: Sanofi bOPV, SII 2 IPV

SUMMARY:
This study is a Phase IV, open, randomized, multi-center, controlled vaccine trial conducted in healthy Latin American infants, utilizing one or two supplemental doses of IPV in children previously vaccinated with 3 doses of bOPV. We will examine the impact of supplemental IPV on stool shedding and humoral immunity, as well as intra-IPV manufacturer comparability, and safety.

DETAILED DESCRIPTION:
The world polio eradication effort is near its goal of reducing the number of new cases of polio to zero. However, final and definitive eradication of the disease will require stopping the use of oral polio vaccines (OPV's) which contain live virus and can rarely revert back to disease producing strains. This period will result in a risk of polio re-emergence as immunity will wane while some vaccine poliovirus will still be circulating. Inactivated polio vaccine (IPV) could potentially play a central role during this process but at present barriers of cost and logistics prevent its routine use in resource limited countries, and concerns exist as to whether IPV provides enough immunity in the intestine to reduce the spread of polioviruses in communities once OPV's are stopped. We plan a multi-center trial in Latin America in which we will administer 1 or 2 doses of IPV to children previously vaccinated with an OPV containing type 1 and 3 poliovirus (bOPV), and then assess the shedding in the stool of a type 2 OPV virus administered later. A decrease in the amount of virus shed compared to children not given IPV would indicate that the IPV boosted intestinal immunity, and would suggest that spread of virus in communities could be reduced using this strategy. We will also measure the impact of supplemental IPV's on antibody formation in the blood, which is a marker of protection of the individual from polio disease. A secondary aim will be to compare the immunogenicity and safety of three IPV's produced by different manufacturers. The overall goal will be to inform policy makers in polio eradication regarding the potential role that one or two doses of IPV might play in the final steps toward polio eradication.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 6 weeks (-7 to +14 days).
2. Healthy without obvious medical conditions that preclude the subject to be in the study as established by the medical history and physical examination.
3. Written informed consent obtained from 1 or 2 parents or legal guardian as per country regulations

Exclusion Criteria:

1. Previous vaccination against poliovirus.
2. Low birth weight (BW <2,500 gm).
3. Multiple pregnancy (twins, triplets, etc.),
4. Any confirmed or suspected immunosuppressive or immunodeficient condition including human immunodeficiency virus (HIV) infection.
5. Family history of congenital or hereditary immunodeficiency.
6. Major congenital defects or serious uncontrolled chronic illness (neurologic, pulmonary, gastrointestinal, hepatic, renal, or endocrine).
7. Known allergy to any component of the study vaccines.
8. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections.
9. Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
10. Acute severe febrile illness at day of vaccination deemed by the Investigator to be a contraindication for vaccination.
11. Member of the subject's household (living in the same house or apartment unit) who has received OPV vaccine in the last 3 months.
12. Subject who, in the opinion of the Investigator or sub-Investigator, is unlikely to comply with the protocol or is inappropriate to be included in the study for the safety or the benefit-risk ratio of the subject.

Min Age: 5 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1420 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in the stool poliovirus excretion after mOPV2 challenge (shedding index) | Within 28 days of mOPV2 challenge
  The basis for calculation of the quantitative shedding index endpoint is to measure the change of viral concentrations shed in stool post-mOPV2 challenge from the baseline timepoint at day 0 to 7, 14, 21 and 28 days as measured from time of mOPV challenge. Quantitative shedding index endpoint will be computed as an area under the viral shedding curve based on these three log10-transformed measurements.
Seroconversion and seroprotection to type 1, 2 and 3 poliovirus | At 6 and 14 weeks, and then before and 1 week after mOPV2 challenge
  The first serologic response endpoint is neutralizing antibody titer defined as the estimated dilution at which 50% neutralizing activity is achieved. The second serologic response endpoint is the binary seroconversion indicator. Seroconversion is considered to be achieved by the time of the subsequent time point if type-specific titers measured at that time are ≥1:8 and > 4-fold over expected levels of maternally-derived antibody computed from the observed titer at baseline assuming an exponential decay with ½ life of 24 days. The third serologic response endpoint of seroprotection is a binary outcome computed from a single antibody titer measurement with seroprotection being achieved if the measured titer is > 1:8.

SECONDARY OUTCOMES:
Comparability of seroconversion and seroprotection from different IPV vaccines | At 6 and 14 weeks, and then before and 1 week after mOPV2 challenge
  To determine whether IPVs from different manufacturers (Sanofi, GSK, SII) are comparable in their ability to induce/boost an antibody response to the 3 poliovirus serotypes in infants vaccinated with 1 or 2 IPV doses after receiving 3 doses of bOPV at 6, 10, and 14 weeks of age
Safety of each vaccine (tOPV, bOPV, mOPV, Sanofi IPV, GSK IPV and SII IPV) and each vaccine schedule | 10 months for each subject
  1. Number of severe adverse events (SAE)throughout the study period
  2. Number of important medical events (IME) as protocol defined: up to 28 days post-vaccination
  3. Number of Local & systemic solicited AEs: 3 days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Edwin J Asturias, MD, Principal Investigator — University of Colorado, Denver; Ricardo Ruttimann, MD, Study Director — Fidec Corporation
Locations (4):
- Centro de Estudios en Infectologia Pediatrica - CEIP, Cali, Cali, Colombia
- Hospital Maternidad Nuestra Señora de la Altagracia, Santo Domingo, Dominican Republic
- Clinica Niño Sano Hospital Roosevelt, Guatemala City, Departamento de Guatemala, Guatemala
- Hospital del Niño de Panama, Panama City, Provincia de Panamá, Panama

REFERENCES:
- [Derived] Lopez-Medina E, Melgar M, Gaensbauer JT, Bandyopadhyay AS, Borate BR, Weldon WC, Ruttimann R, Ward J, Clemens R, Asturias EJ. Inactivated polio vaccines from three different manufacturers have equivalent safety and immunogenicity when given as 1 or 2 additional doses after bivalent OPV: Results from a randomized controlled trial in Latin America. Vaccine. 2017 Jun 16;35(28):3591-3597. doi: 10.1016/j.vaccine.2017.04.041. Epub 2017 Apr 25. PMID 28455172
- [Derived] Asturias EJ, Bandyopadhyay AS, Self S, Rivera L, Saez-Llorens X, Lopez E, Melgar M, Gaensbauer JT, Weldon WC, Oberste MS, Borate BR, Gast C, Clemens R, Orenstein W, O'Ryan G M, Jimeno J, Clemens SA, Ward J, Ruttimann R; Latin American IPV001BMG Study Group. Humoral and intestinal immunity induced by new schedules of bivalent oral poliovirus vaccine and one or two doses of inactivated poliovirus vaccine in Latin American infants: an open-label randomised controlled trial. Lancet. 2016 Jul 9;388(10040):158-69. doi: 10.1016/S0140-6736(16)00703-0. Epub 2016 May 19. PMID 27212429